CLINICAL TRIAL: NCT04261985
Title: A Mobile Phone Based Pilot Intervention to Prevent Obesity in Latino Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alma Guerrero, MD, MPH, Associate Clinical Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R21HD096298-01A1 (NIH); 1R21HD096298-01A1 (NIH)
Record Dates: First submitted 2020-02-03; First posted 2020-02-10 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Childhood Obesity; Parenting; Mobile Phone Use
MeSH Terms: conditions — Pediatric Obesity; Cell Phone Use

STUDY DESIGN:
Intervention Model Description: a prospective control group design
Who Masked: Outcomes Assessor
Masking Description: A research assistant not working on any other aspect of the study, and therefore having no knowledge of whether participants are in the control or intervention group, will measure child and caregiver height and weight. A 2nd research assistant, who is not blinded to participants, will be responsible for making appointments with participants for height and weight measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Phone Obesity Intervention (Active Comparator): Approximately 30 caregiver-child dyads will be randomized into the intervention arm. Every week for 4 weeks, caregivers will receive 4 interactive multi-media phone prompts to support the intervention's targeted topics. Each mobile phone prompt starts with a 140-character text with an embedded link. Clicking on the link navigates caregivers to a web-based application with interactive content that includes images, text, videos, and prompts. Each week, caregivers will share their goal/s, perceived barriers, questions, tips and strategies that may be helpful to other participants. Each week, caregivers will also receive strategies, and individual and group feedback on changing unhealthy behaviors.
  Interventions: Behavioral: healthy weight behaviors supported by web-based mobile phone application
- Control (No Intervention): Approximately 30 caregiver-child dyads will be randomized into the control (no intervention) arm. Every week for 4 weeks, these caregivers will receive 4 interactive multi-media phone prompts around managing common illness in young children (i.e. fever, vomiting, constipation, etc.) Each mobile phone prompt will start with a 140-character text with an embedded link. Clicking on the link navigates caregivers to a web-based application with interactive content that includes images, text, videos, and prompts. Each week, caregivers will share questions and strategies that may be helpful to other participants. Each week, caregivers will also receive tips and group feedback based on group questions.

INTERVENTIONS:
Behavioral: healthy weight behaviors supported by web-based mobile phone application — Chorus is a mobile phone platform that provides texting, a web application, and an online community for mHealth interventions.Content is created using existing templates to insert text, images, pictures, audio, video clips, or any combination of these. Users interface with Chorus by clicking a hyperlink embedded in a text message sent to their phone to then access web-based interactions via prompts and clicks. Content was created in English and Spanish.
  Arms: Mobile Phone Obesity Intervention

SUMMARY:
To pilot a stand-alone mobile phone intervention with Latino caregivers of 2- to 5-year olds, using a prospective control group design, to assess feasibility and preliminary effect sizes on children's BMI changes (primary outcome) and dietary and physical activity changes (secondary outcomes) at 6 months post-baseline, in preparation for a larger randomized trial to evaluate the intervention's efficacy.

DETAILED DESCRIPTION:
The investigators will pilot an mHealth intervention using a prospective control group design with 66 caregiver-child dyads (33 intervention and 33 comparison) recruited from two community based agencies in East Los Angeles. Fidelity and feasibility will be assessed. Pre- and post- intervention data (child dietary, physical activity, and media viewing behaviors and BMI z-scores) will be collected to estimate preliminary effect sizes and standard deviations. The mHealth intervention has been informed by a previous feasibility study and focus groups with Latino caregivers of 2- to 5-year old children. This mHealth childhood obesity intervention specifically targets Latino mothers, fathers, and grandmothers of 2- to 5-year olds. The intervention focuses on parenting skills, dietary, physical activity, and media-viewing behaviors consistent with American Academy of Pediatrics guidelines.

ELIGIBILITY:
Inclusion Criteria:

* adult male or female caregiver
* self-identifies as an individual of Latino descent
* has a child or grandchild 2-5 years of age (relationship does not have to be biological but caregiver is a legal guardian)
* lives with or cares for child/grandchild at least 20 hours/week
* is fluent in English or Spanish
* has the ability to participate in the mHealth intervention (ability determined by using a Subject Comprehension and Participation Assessment Tool)
* agrees to complete baseline, 1-, and 6-month post-baseline surveys and have adult and child height and weight measured.

Exclusion Criteria:

* child has a failure to thrive diagnosis
* medical complications associated with their weight status such as Prader-Willi Syndrome

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study set out to enroll 60 parent-child dyads. Every parent-child dyad consists of one child between 2-years old and 5-years old and the child's primary caregiver. We, therefore, set out to enroll a total of 120 participants (60 children and 60 caregivers).
Groups:
- Mobile Phone Obesity Intervention: Caregiver-child dyads will be recruited from two early childhood education centers in East Los Angeles. Approximately 30 caregiver-child dyads will be randomized into the intervention arm. Every week for 4 weeks, caregivers will receive 4 interactive multi-media phone prompts to support the intervention's targeted topics. Each mobile phone prompt starts with a 140-character text with an embedded link. Clicking on the link navigates caregivers to a web-based application with interactive content that includes images, text, videos, and prompts. Each week, caregivers will share their goal/s, perceived barriers, questions, tips and strategies that may be helpful to other participants. Each week, caregivers will also receive strategies, and individual and group feedback on changing unhealthy behaviors. The content shared by caregivers are summarized by a team research assistant and sent back to participants at the end of every week.
  healthy weight behaviors supported by web-based mobile phone application: Chorus is a mobile phone platform that provides texting, a web application, and an online community for mHealth interventions.Content is created using existing templates to insert text, images, pictures, audio, video clips, or any combination of these. Users interface with Chorus by clicking a hyperlink embedded in a text message sent to their phone to then access web-based interactions via prompts and clicks. Content is available in English and Spanish.
- Control: Caregiver-child dyads will be recruited from two early childhood education centers in East Los Angeles. Approximately 30 caregiver-child dyads will be randomized into the control (no intervention) arm. Every week for 4 weeks, these caregivers will receive 4 interactive multi-media phone prompts around managing common illness in young children (i.e. fever, vomiting, constipation, etc.) Each mobile phone prompt will start with a 140-character text with an embedded link. Clicking on the link navigates caregivers to a web-based application with interactive content that includes images, text, videos, and prompts. Each week, caregivers will share questions and strategies that may be helpful to other participants. Each week, caregivers will also receive tips and group feedback based on group questions. The content shared by caregivers will be summarized by a team research assistant and sent back to participants at the end of every week.
Period: Baseline
Arm/Group | Mobile Phone Obesity Intervention | Control
Started | 54 | 64
Completed | 54 | 64
Not Completed | 0 | 0
Period: 6-month Follow-up
Arm/Group | Mobile Phone Obesity Intervention | Control
Started | 54 | 64
Completed | 52 | 62
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Phone Obesity Intervention | Control | Total
Number analyzed (Participants) | 54 | 64 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 32 | 59
  Between 18 and 65 years | 27 | 32 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — child and caregiver age in years Population: Study included children and caregivers.
  years
    Children: number analyzed (Participants) | 27 | 32 | 59
    Children | 4.0 (0.9) | 4.1 (0.8) | 4.0 (0.9)
    Caregivers: number analyzed (Participants) | 27 | 32 | 59
    Caregivers | 32.3 (8.6) | 35.2 (7.6) | 34 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The first row is the % of male and females of children in the study, the second row is % of male and females of caregivers in study
  Participants
    children: number analyzed (Participants) | 27 | 32 | 59
    children: Female | 15 | 16 | 31
    children: Male | 12 | 16 | 28
    caregivers: number analyzed (Participants) | 27 | 32 | 59
    caregivers: Female | 26 | 29 | 55
    caregivers: Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The first row relates to the % of Latino children and the second row is related to % of Latino caregivers
  Participants
    Children: number analyzed (Participants) | 27 | 32 | 59
    Children: Hispanic or Latino | 27 | 32 | 59
    Children: Not Hispanic or Latino | 0 | 0 | 0
    Children: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 27 | 32 | 59
    Caregivers: Hispanic or Latino | 27 | 32 | 59
    Caregivers: Not Hispanic or Latino | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 64 | 118
pounds [Mean (Standard Deviation); unit: lbs] — Population: The first row are results for children and the second row for caregivers.
  lbs
    Children: number analyzed (Participants) | 27 | 32 | 59
    Children | 41.1 (7.9) | 40.4 (7.3) | 40.6 (7.6)
    Caregivers: number analyzed (Participants) | 27 | 32 | 59
    Caregivers | 171 (35.6) | 176 (35.6) | 173 (33.1)

OUTCOME MEASURES:

1. Primary Outcome: Child Weight
Description: Child pounds measured using participant weight measured on a digital scale (calibrated with 5kg weight before each measurement) to the nearest 0.1 pounds
Time Frame: 6-months post baseline
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Mobile Phone Obesity Intervention | Control
Number analyzed (Participants) | 26 | 31
lbs | 45.6 (9.7) | 44.9 (8.6)

2. Secondary Outcome: Caregiver Weight in Pounds
Description: Caregiver pounds measured using participant weight measured on a digital scale (calibrated with 5kg weight before each measurement) to the nearest 0.1 pounds
Time Frame: 6-months post-intervention
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Mobile Phone Obesity Intervention | Control
Number analyzed (Participants) | 26 | 31
pounds | 176.9 (35.1) | 178.3 (32.9)

ADVERSE EVENTS:
Time Frame: No adverse events occurred through study completion, on average 10 months.
Arm/Group | Mobile Phone Obesity Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/64
Other Adverse Events (participants affected / at risk) | 0/54 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT04261985/Prot_SAP_000.pdf